CLINICAL TRIAL: NCT02418117
Title: Accuracy of Computer Guided Implant Surgery With the Use of R2Gate Stereolitographic Template
Brief Title: Accuracy of Computer Guided Implant Surgery
Acronym: STIMPLANTSRG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia Dent Srl (Other)
Collaborators: Carol Davila University of Medicine and Pharmacy (Other); MEGAGEN DENTAL IMPLANT ROMANIA (Unknown)
Responsible Party: Principal Investigator, Corina Marilena Cristache, Dr Corina Marilena Cristache, DMD, PhD, senior lecturer, Concordia Dent Srl
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 613/15
Record Dates: First submitted 2015-04-09; First posted 2015-04-16 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Jaw, Edentulous
Keywords: Stereolitographic guide; flapless surgery; dental implants
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereolitographic template's accuracy (Experimental): Evaluating the accuracy of stereolitographic template comparing the final implant insertion to the planned implant position at coronal and apical level
  Interventions: Other: Stereolitographic template

INTERVENTIONS:
Other: Stereolitographic template — Flapless (atraumatic) dental implants insertion with the aid of a stereolitographic template.

SUMMARY:
The investigators' aim is to evaluate the accuracy of the stereolitographic template comparing the final implant insertion to the planned implant position at coronal and apical level.

Clinical relevance:

* To identify factors influencing the surgical template imprecision.
* To overcome risk factors for surgical template imprecision.
* To suggest improvements for highly accuracy of the surgical template especially for immediate loading and avoiding the injury of anatomical structures.

DETAILED DESCRIPTION:
Initial examination, panoramic radiograph to be performed and impression for stone models to be taken to all enrolled patients. For diagnosis accuracy, impression of the surgical site and the opposite arch is mandatory.

For fully edentulous and extensive edentulous subjects - Class III and IV according to the American College of Prosthodontists - ACP - a visible light cure record bases with occlusal rims will be manufactured for bite registration.

CBCT will be taken with a R2 tray filled with impression material or with record basis in centric relation (CR).

CBCT will be performed using same CT machine with a specific setup and alignment to allow accuracy and reproducibility.

A series of axially sliced image data will be obtained and exported to a personal computer in DICOM (Digital Imaging and Communications in Medicine) format.

Models, occlusal rims and R2 trays will be scanned and imported as STL (Stereo Lithography) files.

On the scan models, a virtual wax-up will be designed with the use of 3Shape CAD (Computer Aided Design) software and saved as STL file.

Matching CT and models scan data DICOM files obtained from CBCT and STL files will be imported in a treatment plan software R2GATE version 1.0.3 (Megagen Implant, Korea) and implant insertion will be planned according to the final restoration and bone anatomy.

AnyRidge Megagen implants will be used with length and diameters required by the clinical cases.

A stereolitographic template manufactured by DDX Europa, after final decision of treatment plan, will be used for dental implants insertion using a minimally invasive flapless approach.

To assess accuracy of the surgical template, a new CBCT with specific set-up and alignment after implant insertion will be performed.

Matching post-op CT with the planed position of the implants will be performed using the R2GATE software and measurements between the location of implants on CT at the time of planning and after implantation will be made at the coronal and apical levels to determine the distance between the implant and the planned position buccal, oral, mesial and distal by two independent researchers. Angulation between the implant position and the planned position at coronal and apical level will be also measured.

Statistical analysis will be performed. Teeth supported, mucosal supported and teeth-mucosal supported surgical stereolitographic template will be analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

* fully or partially edentulous patients,
* good general healty with no contraindications for implant surgery,
* acceptance of dental implant treatment,
* acceptance of at least 2 CBCT (one at treatment planning and one after surgery)

Exclusion Criteria:

* limited bone volume with stadial bone graft requirement,
* limited mouth opening (imposible to use the surgical stent),
* parkinson desease (imposible to perform an accurate CBCT)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Measurements of accuracy after implants placement at coronal and apical level | average 10 days
  Measurements between the location of implants on CT at the time of planning and after implantation will be made at the coronal and apical levels to determine the distance between the implant and the planned position buccal, oral, mesial and distal.

CONTACTS AND LOCATIONS:
Overall Officials: CORINA MARILENA I CRISTACHE, DMD, PhD, Principal Investigator — Carol Davila University of Medicine and Pharmacy
Locations (1):
- Concordia Dent Clinic, Bucharest, Romania

REFERENCES:
- [Background] Vasak C, Kohal RJ, Lettner S, Rohner D, Zechner W. Clinical and radiological evaluation of a template-guided (NobelGuide) treatment concept. Clin Oral Implants Res. 2014 Jan;25(1):116-23. doi: 10.1111/clr.12038. Epub 2012 Sep 18. PMID 22984962
- [Background] Yatzkair G, Cheng A, Brodie S, Raviv E, Boyan BD, Schwartz Z. Accuracy of computer-guided implantation in a human cadaver model. Clin Oral Implants Res. 2015 Oct;26(10):1143-9. doi: 10.1111/clr.12482. Epub 2014 Sep 15. PMID 25220954
- [Background] Beretta M, Poli PP, Maiorana C. Accuracy of computer-aided template-guided oral implant placement: a prospective clinical study. J Periodontal Implant Sci. 2014 Aug;44(4):184-93. doi: 10.5051/jpis.2014.44.4.184. Epub 2014 Aug 28. PMID 25177520
- [Background] Van Assche N, Vercruyssen M, Coucke W, Teughels W, Jacobs R, Quirynen M. Accuracy of computer-aided implant placement. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:112-23. doi: 10.1111/j.1600-0501.2012.02552.x. PMID 23062136